CLINICAL TRIAL: NCT01453348
Title: A Phase 3b, Randomized, Open-Label Study to Evaluate the Safety and Immunogenicity of Combined Hepatitis A/B Vaccine When Administered Concomitantly With Novartis Meningococcal ACWY Conjugate Vaccine in Healthy Adults
Brief Title: Study to Evaluate the Safety and Immunogenicity of Combined Hepatitis A/B Vaccine With MenACWY-CRM Conjugate Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V59_53; 2011-001333-17 (EudraCT Number)
Record Dates: First submitted 2011-10-03; First posted 2011-10-17 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Meningococcal Disease; Meningococcal Meningitis; Hepatitis A; Hepatitis B
Keywords: meningococcal; conjugate; vaccine; adults
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal; Hepatitis A; Hepatitis B | interventions — MenACWY-CRM vaccine; Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): This group will receive Inactivated hepatitis A and recombinant hepatitis B or 'Combined inactivated hepatitis A & recombinant hepatitis B vaccine' alone on the different visits.
  Interventions: Biological: Combined inactivated hepatitis A & recombinant hepatitis B; Biological: Recombinant hepatitis B vaccine; Biological: Inactivated hepatitis A vaccine
- Group 2 (Active Comparator): This group will receive Inactivated hepatitis A vaccine and recombinant hepatitis B Vaccine or 'Combined inactivated hepatitis A & recombinant hepatitis B vaccine' concomitantly with MenACWY-CRM.
  Interventions: Biological: MenACWY-CRM; Biological: Combined inactivated hepatitis A & recombinant hepatitis B; Biological: Recombinant hepatitis B vaccine; Biological: Inactivated hepatitis A vaccine
- Group 3 (Active Comparator): This group will receive only MenACWY-CRM.
  Interventions: Biological: MenACWY-CRM

INTERVENTIONS:
Biological: MenACWY-CRM — Novartis meningococcal ACWY conjugate vaccine will be administered intramuscularly (IM) on day 1.
  Arms: Group 2; Group 3
Biological: Combined inactivated hepatitis A & recombinant hepatitis B — Combined inactivated hepatitis A and recombinant hepatitis B vaccine will be administered by IM on days 1, 8 & 29 for subjects unprimed with hepatitis A and B; and a single booster injection on day 1 for primed subjects.
  Arms: Group 1; Group 2
Biological: Recombinant hepatitis B vaccine — Recombinant hepatitis B vaccine will be administered intramuscularly on days 8 and 29
  Arms: Group 1; Group 2
Biological: Inactivated hepatitis A vaccine — Inactivated hepatitis A will be administered intramuscularly on days 8 and 29.
  Arms: Group 1; Group 2

SUMMARY:
This study compares the safety and immunogenicity profile of combined hepatitis A/B vaccine given alone or concomitantly with MenACWY-CRM to healthy adults.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible for enrollment in this study were female and male subjects who had shown to be healthy and who were:

1. Between 18 and 64 years of age inclusive and who had given their written informed consent;
2. Available for all visits and telephone calls scheduled for the study;
3. In good health as determined by medical history, physical examination and clinical judgment of the investigator;
4. For female subjects, had a negative urine pregnancy test.

Exclusion Criteria:

Individuals not eligible to be enrolled in the study were those:

1. Who were breastfeeding.
2. Who had a previous personal history of Neisseria meningitidis, hepatitis A or hepatitis B infection.
3. Who received previous immunization with any meningococcal vaccine.
4. Who received previous hepatitis A and/or B vaccination, determined by history (interview of the subject) and/or by review of his or her vaccination card, if less than 5 years have elapsed since vaccination.
5. Who received investigational agents or vaccines within 30 days prior to enrollment or who expected to receive an investigational agent or vaccine prior to completion of the study.
6. Who received live licensed vaccines within 30 days and inactive vaccine within 15 days prior to enrollment or for whom receipt of a licensed vaccine was anticipated during the study period (Exception: Influenza vaccine might have been administered up to 15 days prior to each study immunization and no less than 15 days after each study immunization).
7. Who experienced, within the 7 days prior to enrollment, significant acute infection (for example requiring systemic antibiotic treatment or antiviral therapy) or had experienced fever (defined as body temperature ≥ 38°C) within 3 days prior to enrollment.
8. Who had any serious acute, chronic or progressive disease such as:

   * History of cancer
   * Complicated diabetes mellitus
   * Advanced arteriosclerotic disease
   * Autoimmune disease
   * HIV infection or AIDS
   * Blood dyscrasias
   * Congestive heart failure
   * Renal failure
   * Severe malnutrition (Note: Subjects with mild asthma were eligible for enrollment. Subjects with moderate or severe asthma requiring routine use of inhaled or systemic corticosteroids were not eligible for enrollment).
9. Who had epilepsy, any progressive neurological disease or history of Guillain-Barre syndrome.
10. Who had a history of anaphylaxis, serious vaccine reactions, or allergy to any vaccine component, including but not limited to latex allergy and antibiotic allergy.
11. Who had a known or suspected impairment/alteration of immune function, either congenital or acquired or resulting from (for example):

    * Receipt of immunosuppressive therapy within 30 days prior to enrollment (systemic corticosteroids administered for more than 5 days, or in a daily dose > 1 mg/kg/day prednisone or equivalent during any of 30 days prior to enrollment, or cancer chemotherapy);
    * Receipt of immunostimulants;
    * Receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within 90 days prior to enrollment and for the full length of the study.
12. Who were known to have a bleeding diathesis, or any condition that might have been associated with a prolonged bleeding time.
13. Who had any condition that, in the opinion of the investigator, might have interfered with the evaluation of the study objectives.
14. Who were part of the study personnel or close family members of those conducting this study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 252 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (4):
- Germany (4):
  - 03, Novartis Investigational Site, Berlin
  - 02, Novartis Investigational Site, Hamburg
  - 01, Novartis Investigational Site, München
  - 04, Novartis Investigational Site, Rostock

REFERENCES:
- [Derived] Alberer M, Burchard G, Jelinek T, Reisinger EC, Meyer S, Forleo-Neto E, Dagnew AF, Arora AK. Immunogenicity and safety of concomitant administration of a combined hepatitis A/B vaccine and a quadrivalent meningococcal conjugate vaccine in healthy adults. J Travel Med. 2015 Mar-Apr;22(2):105-14. doi: 10.1111/jtm.12180. Epub 2014 Dec 7. PMID 25483566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at four centers in Germany.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- HepA/B: Subjects ≥ 18 to ≤ 64 years of age who were not previously primed with hepatitis A and B vaccine received three doses of combined hepatitis A/B vaccine; subjects who were previously primed with combined hepatitis A/B received one booster dose; subjects who were previously primed with monovalent hepatitis B vaccine received one dose of combined hepatitis A/B vaccine on day 1 (hepatitis B vaccine booster; first dose of hepatitis A vaccine on an accelerated schedule), followed by two doses of monovalent hepatitis A vaccine; subjects who were previously primed with hepatitis A vaccine received one dose of combined hepatitis A/B vaccine on day 1 (hepatitis A vaccine booster; first dose of hepatitis B vaccine on an accelerated schedule), followed by two doses of monovalent hepatitis B vaccine.
- HepA/B+MenACWY-CRM: Subjects ≥ 18 to ≤ 64 years of age who were not previously primed with hepatitis A and B vaccine received three doses of combined hepatitis A/B vaccine; subjects who were previously primed with combined hepatitis A/B received one booster dose; subjects who were previously primed with monovalent hepatitis B vaccine received one dose of combined hepatitis A/B vaccine on day 1 (hepatitis B vaccine booster; first dose of hepatitis A vaccine on an accelerated schedule), followed by two doses of monovalent hepatitis A vaccine; subjects who were previously primed with hepatitis A vaccine received one dose of combined hepatitis A/B vaccine on day 1 (hepatitis A vaccine booster; first dose of hepatitis B vaccine on an accelerated schedule), followed by two doses of monovalent hepatitis B vaccine; all the subjects concomitantly received one dose of MenACWY-CRM conjugate vaccine.
- MenACWY-CRM: Subjects ≥ 18 to ≤ 64 years of age who received one dose of MenACWY-CRM conjugate vaccine.
Period: Overall Study
Arm/Group | HepA/B | HepA/B+MenACWY-CRM | MenACWY-CRM
Started | 84 | 84 | 84
Completed | 83 | 83 | 83
Not Completed | 1 | 1 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HepA/B | HepA/B+MenACWY-CRM | MenACWY-CRM | Total
Number analyzed (Participants) | 84 | 84 | 84 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (12.3) | 39.9 (12.6) | 39.7 (11.0) | 39.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 40 | 50 | 135
  Male | 39 | 44 | 34 | 117

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean antiHAV and antiHBV Concentrations (GMCs), 28 Days After Primary and Booster Vaccination
Description: Assessment was made to demonstrate the non-inferiority of hepatitis A/B vaccine with MenACWY-CRM as compared to hepatitis A/B vaccine without MenACWY-CRM, as measured by geometric mean concentrations on day 57 in previously unvaccinated subjects or on day 29 after a booster dose in previously vaccinated subjects.
Time Frame: Day 57 (previously unprimed subjects) day 29 (previously primed subjects) postvaccination.
Population: Analysis was done on Per Protocol (PP) population who provided evaluable serum samples and whose assay results were available at the relevant time points, and had no major protocol deviations
Measure: Geometric Mean (95% Confidence Interval); unit: Concentrations (mIU/mL)
Groups:
- HepA/B+MenACWY-CRM: Subjects ≥ 18 to ≤ 64 years of age who were not previously primed with hepatitis A and B vaccine received three doses of combined hepatitis A/B vaccine; subjects who were previously primed with combined hepatitis A/B received one booster dose; subjects who were previously primed with monovalent hepatitis B vaccine received one dose of combined hepatitis A/B vaccine on day 1 (hepatitis B vaccine booster; first dose of hepatitis A vaccine on an accelerated schedule), followed by two doses of monovalent hepatitis A vaccine ; subjects who were previously primed with hepatitis A vaccine received one dose of combined hepatitis A/B vaccine on day 1 (hepatitis A vaccine booster; first dose of hepatitis B vaccine on an accelerated schedule), followed by two doses of monovalent hepatitis B vaccine; all the subjects concomitantly received one dose of MenACWY-CRM conjugate vaccine.
Arm/Group | HepA/B+MenACWY-CRM | HepA/B
Number analyzed (Participants) | 78 | 78
Concentrations (mIU/mL)
  Prevaccination AntiHAV | 48 [27 to 85] | 30 [17 to 54]
  28 days after primary or booster AntiHAV | 786 [591 to 1046] | 884 [664 to 1176]
  Prevaccination AntiHBV (N=78, 76) | 22 [12 to 39] | 31 [17 to 57]
  28 days after primary or booster AntiHBV (N=78,76) | 844 [513 to 1387] | 711 [429 to 1179]
Statistical Analysis 1: Comparison: HepA/B+MenACWY-CRM vs HepA/B; The primary criterion for immunogenicity was that the lower-limit of the two-sided 95% Confidence Interval (CI) on the ratio of Enzyme-linked Immunosorbent Assay (ELISA) GMCs (Hep A/B + MenACWY-CRM to Hep A/B) is below or equal to 0.5; Test type: Non-Inferiority or Equivalence — (GMC anti-HAV + MenACWY-CRM / GMC anti-HAV); ANCOVA — The testing was done by assessing the confidence interval of the ratio; The Analysis of variance (ANCOVA) model included vaccine group and center as factors, age as covariate and was adjusted for baseline; Ratio of GMC = 0.89, 95% CI 2-sided [0.6 to 1.32]
Statistical Analysis 2: Comparison: HepA/B+MenACWY-CRM vs HepA/B; The primary criterion for immunogenicity was that the the lower-limit of the two-sided 95% CI on the ratio of ELISA GMCs (Hep A/B + MenACWY-CRM to Hep A/B) is below or equal to 0.5; Test type: Non-Inferiority or Equivalence — (GMC anti-HBsAg + MenACWY-CRM / GMC anti-HBsAg); ANCOVA — The testing was done by assessing the confidence interval of the ratio; The ANCOVA model included vaccines group and center as factors, age as covariate and was adjusted for baseline; Ratio of GMC = 1.19, 95% CI 2-sided [0.59 to 2.37]

2. Secondary Outcome: Percentages of Subjects With antiHAV and antiHBsAg Antibodies Concentrations Above Seroprotection Level 28 Days After Primary or Booster Vaccination
Description: Immunogenicity was assessed as the percentages of subjects with anti-HAV concentration ≥20 mIU/mL and anti- HBsAg antibody concentration ≥10 mIU/mL, 28 days after primary or booster vaccination.
Time Frame: 28 days post primary or booster vaccination.
Population: Analysis was done on modified intention-to-treat (MITT) population- subjects who provided evaluable serum samples whose assay results are available for at least one antigen on visit day 1 and a post baseline visit.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | HepA/B+MenACWY-CRM | HepA/B
Number analyzed (Participants) | 83 | 82
percentage of subjects
  AntiHAV antibody concentration ≥20mIU/mL (Day 1) | 42 [31 to 54] | 33 [23 to 44]
  28 days after primary/booster AntiHAV | 96 [90 to 99] | 99 [93 to 100]
  AntiHBsAg antibody concentration ≥10mIU/mL (Day 1) | 47 [36 to 58] | 44 [33 to 55]
  28 days after primary/booster AntiHBV | 75 [64 to 84] | 80 [70 to 88]

3. Secondary Outcome: Percentages of Subjects With Seroresponse Against N Meningitidis A, C, W and Y Serogroups at Day 29
Description: Immunogenicity was assessed as the seroresponse rates for meningococcal serogroups A, C, W and Y elicited by MenACWY-CRM on day 29 when given concomitantly with combined hepatitis A/B vaccine or given alone.
  For a subject with a baseline hSBA titer < 1:4, seroresponse is defined as a postvaccination hSBA titer ≥1:8; for a subject with a baseline hSBA titer ≥ 1:4, seroresponse is defined as a postvaccination hSBA titer of at least 4 times the baseline.
Time Frame: 28 days postvaccination (day 29).
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | HepA/B+MenACWY-CRM | MenACWY-CRM
Number analyzed (Participants) | 83 | 83
percentage of subjects
  MenA-hSBA Overall Seroresponse (N=83, 82) | 71 [60 to 81] | 65 [53 to 75]
  MenC-hSBA Overall Seroresponse | 66 [55 to 76] | 59 [48 to 70]
  MenW-hSBA Overall Seroresponse (N=83, 82) | 40 [29 to 51] | 34 [24 to 45]
  MenY-hSBA Overall Seroresponse | 70 [59 to 79] | 64 [53 to 74]

4. Secondary Outcome: hSBA GMTs Assay Titers Against N Meningitidis A, C, W and Y Serogroups at Day 29
Description: Immunogenicity was assessed in terms of geometric mean titers (GMTs) of antibodies to meningococcal serogroups A, C, W and Y on day 29 when given concomitantly with combined hepatitis A/B vaccine or given alone.
Time Frame: 28 days post vaccination (day 29).
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | HepA/B+MenACWY-CRM | MenACWY-CRM
Number analyzed (Participants) | 84 | 84
Titers
  Men A Human Complement SBA; Day 1 (N= 84, 84) | 2.68 [2.27 to 3.17] | 2.71 [2.29 to 3.2]
  Men A Human Complement SBA; Day 29 (N=83, 82) | 43 [27 to 67] | 36 [23 to 58]
  Men C Human Complement SBA; Day 1 (N= 84, 84) | 7.39 [5.49 to 9.94] | 6.35 [4.71 to 8.57]
  Men C Human Complement SBA; Day 29 (N=83, 83) | 75 [50 to 112] | 56 [37 to 83]
  Men W Human Complement SBA; Day 1 (N=84, 83) | 30 [21 to 42] | 31 [22 to 45]
  Men W Human Complement SBA; Day 29 (N=83, 83) | 110 [84 to 145] | 109 [82 to 144]
  Men Y Human Complement SBA; Day 1 (N= 84, 84) | 6.63 [5.06 to 8.68] | 5.56 [4.23 to 7.3]
  Men Y Human Complement SBA; Day 29 (N=83, 83) | 78 [55 to 111] | 62 [44 to 89]

5. Secondary Outcome: Percentages of Subjects With Unsolicited Adverse Events (AEs)
Description: Safety was assessed in terms of percentage of all spontaneously reported AEs collected from the time the subject signed the informed consent form (day 1), until the subject stopped study participation (day 57).
Time Frame: Day 1 to day 57.
Population: Analysis was done on safety set- subjects who provided any post-baseline safety data.
Measure: Number; unit: percentage of subjects
Arm/Group | HepA/B | HepA/B+MenACWY-CRM | MenACWY-CRM
Number analyzed (Participants) | 84 | 85 | 83
percentage of subjects
  Any AE | 43 | 39 | 36
  Atleast possibly related AE | 23 | 27 | 17
  Any SAE | 1 | 0 | 1
  AE leading to withdrawal | 0 | 1 | 1
  Death | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 1 to day 57.
Description: Safety was assessed in terms of percentages of all Serious AEs collected from the time the subject signed the informed consent form until he/she stopped study participation.One subject randomized to receive MenACWY-CRM, received HepA/B+MenACWY-CRM vaccine, instead. The safety set included 85 subjects for HepA/B+MenACWY group and 83 for MenACWY.
Groups:
- HepA/B: Subject ≥ 18 to ≤ 64 years of age who were not previously primed with hepatitis A and B vaccine received three doses of combined hepatitis A/B vaccine; subjects who were previously primed with combined hepatitis A/B received one booster dose; subjects who were previously primed with monovalent hepatitis B vaccine received one dose of combined hepatitis A/B vaccine on day 1 (hepatitis B vaccine booster; first dose of hepatitis A vaccine on an accelerated schedule), followed by two doses of monovalent hepatitis A vaccine; subjects who were previously primed with hepatitis A vaccine received one dose of combined hepatitis A/B vaccine on day 1 (hepatitis A vaccine booster; first dose of hepatitis B vaccine on an accelerated schedule), followed by two doses of monovalent hepatitis B vaccine.
- HepA/B+ACWY: Subject ≥ 18 to ≤ 64 years of age who were not previously primed with hepatitis A and B vaccine received three doses of combined hepatitis A/B vaccine; subjects who were previously primed with combined hepatitis A/B received one booster dose; subjects who were previously primed with monovalent hepatitis B vaccine received one dose of combined hepatitis A/B vaccine on day 1 (hepatitis B vaccine booster; first dose of hepatitis A vaccine on an accelerated schedule), followed by two doses of monovalent hepatitis A vaccine; subjects who were previously primed with hepatitis A vaccine received one dose of combined hepatitis A/B vaccine on day 1 (hepatitis A vaccine booster; first dose of hepatitis B vaccine on an accelerated schedule), followed by two doses of monovalent hepatitis B vaccine; all the subjects concomitantly received one dose of MenACWY-CRM conjugate vaccine.
- ACWY: Subject ≥ 18 to ≤ 64 years of age who received one dose of MenACWY-CRM conjugate vaccine.
Arm/Group | HepA/B | HepA/B+ACWY | ACWY
Serious Adverse Events (participants affected / at risk) | 1/84 | 0/85 | 1/83
Other Adverse Events (participants affected / at risk) | 25/84 | 21/85 | 12/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HepA/B (N=84) | HepA/B+ACWY (N=85) | ACWY (N=83)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
COMPLETED SUICIDE (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HepA/B (N=84) | HepA/B+ACWY (N=85) | ACWY (N=83)
FATIGUE (General disorders) | 2 | 6 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 2 | 1 | 5
INJECTION SITE PAIN (General disorders) | 4 | 5 | 1
NASOPHARYNGITIS (Infections and infestations) | 6 | 9 | 5
HEADACHE (Nervous system disorders) | 15 | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No